CLINICAL TRIAL: NCT05239247
Title: Effects of Eldoa Versus Meckenzie Exercise on Non-specific Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muniba Shamshad
Record Dates: First submitted 2022-02-01; First posted 2022-02-14 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mckenzie extension exercise (Experimental)
  Interventions: Other: Mckenzie extension exercise
- Eldoa stretch technique (Experimental)
  Interventions: Other: Eldoa stretch technique

INTERVENTIONS:
Other: Mckenzie extension exercise — Hot pack applied on lumbar region for (ten minute). Mckenzie extension exercise performed 02 sets of 05 repetitions with 45 second hold and 15 sec rest between each set once a day.
  TENS is applied on lumbar region for (ten minutes).
  Arms: Mckenzie extension exercise
Other: Eldoa stretch technique — Hot pack applied on lumbar region for (ten minute). Eldoa stretch performed 02 sets of 05 repetitions with 45 second hold and 15 second rest between each set once a day.
  TENS is applied on lumbar region for (ten minutes).
  Arms: Eldoa stretch technique

SUMMARY:
To determine the effects of Eldoa and Mckenzie exercises in posture. To determine the effects of Eldoa and Mckenzie exercises in ROM.

DETAILED DESCRIPTION:
To determine the effects of Eldoa and Mckenzie exercises in pain. To determine the effects of Eldoa and Mckenzie exercises in Quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Gender (Female)
* Age (40-69)
* NPRS (Grade <3)
* Chronic pain (more than or equal to 3 months)
* Restricted ROM
* Lumbar straightening

Exclusion Criteria:

* Any other orthopedic or neurological condition of hip or lumbar spine.
* sign and symptoms of lower motor neuron disease.
* Current use of medication prescribed for pain.
* Radiculopathy.
* malignancy.
* Fracture.
* Lumbar trauma.
* Disc pathology

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female age between 40 -69
Enrollment: 48 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
lumbar ROM by inclinometer. | 12 days
  Flexion 60 Extension 25 Left Lat Flex 25 Right Lat Flex 25
Lumbar Posture by flexicurve ruler. | 12 days
  Excessive lordosis (EL) is over 75°, normal lordosis (NL) is 40°, hypo-lordosis (HL) is in the 20°

SECONDARY OUTCOMES:
pain on Numeric pain rating scale. | 12 days
  Changes from baseline, Pain was measured through Numeric pain rating scale.It comprises of a continuous scale of 10cm line.0 to 1 represent no pain, 1 to 3 represent mild pain ,4 to 6 represent moderate pain, 7 to 10 represent severe pain.
functional outcome by Oswestry low back pain disability questionnaire. | 12 days
  0% to 20%: minimal disability: The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise. 21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required. 81%-100%:These patients are either bed-bound or exaggerating their symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rawal General And Dental Hospital, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No